CLINICAL TRIAL: NCT00841061
Title: Breast Feeding and Iron: Comparison of Cereals Fortified With Different Forms of Iron
Brief Title: Cereals as a Source of Iron for Breastfed Infants
Acronym: Bfe03B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health (NIH) (NIH)
Responsible Party: Dr. Ekhard E. Ziegler, University of Iowa
Organization: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B530500; HD40315-01
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-01

CONDITIONS: Iron Deficiency
MeSH Terms: conditions — Iron Deficiencies | interventions — ferrous fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cereal L (Active Comparator): Rice cereal with electrolytic iron
  Interventions: Dietary Supplement: electrolytic iron
- Cereal M (Active Comparator): Rice cereal with ferrous fumarate
  Interventions: Dietary Supplement: ferrous fumarate

INTERVENTIONS:
Dietary Supplement: electrolytic iron — 1/4 a cup of cereal fortified with electrolytic iron per day between the ages of 112 days and 280 days of age
  Arms: Cereal L
Dietary Supplement: ferrous fumarate — 1/4 cup of cereal fortified with ferrous fumarate to be fed per day between ages of 112 days and 280 days of age
  Arms: Cereal M

SUMMARY:
The purpose of this research study is to determine whether the type of iron in infant cereals makes a differance in how well the cereal helps infants remain free of iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* exclusively breastfed
* birth weight between 2500 and 4200g
* gestational age >36 weeks

Exclusion Criteria:

* supplementing formula
* no iron drops

Ages: 28 Days to 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 111 (Actual)
Dates: Start 2003-07; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
plasma ferritin | 280 days

SECONDARY OUTCOMES:
hemoglobin | 280

CONTACTS AND LOCATIONS:
Overall Officials: Ekhard E Ziegler, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Ziegler EE, Fomon SJ, Nelson SE, Jeter JM, Theuer RC. Dry cereals fortified with electrolytic iron or ferrous fumarate are equally effective in breast-fed infants. J Nutr. 2011 Feb;141(2):243-8. doi: 10.3945/jn.110.127266. Epub 2010 Dec 22. PMID 21178077